CLINICAL TRIAL: NCT05718908
Title: Pilot Study of a Cohort of Patients Affected by Fibromyalgia for Symptomatic Improvement by Means of a Food Supplement
Brief Title: Study of the Symptomatic Improvement in Patients With Fibromyalgia by Means of a Food Supplement
Acronym: FIBROFIN
Status: Completed | Type: Observational
Sponsor: Arafarma Group, S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: ARA-OBS/FIB-2021-01
Record Dates: First submitted 2022-11-28; First posted 2023-02-08 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Dietary Supplements

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fibromyalgia patients: All patients will be administered with one sachet of food supplement (FibrofixPlus®) per day, for 8 weeks.
  Interventions: Dietary Supplement: Food supplement

INTERVENTIONS:
Dietary Supplement: Food supplement — FibrofixPlus® is an authorized food supplement.

SUMMARY:
Fibromyalgia is a syndrome (set of symptoms) of unknown etiology and characterized by diffuse musculoskeletal pain and chronic fatigue. In addition, other symptoms such as cognitive alterations, sleep rhythm disturbances, psychiatric syndromes such as anxiety, depression, etc. Other very characteristic symptoms are hyperalgesia (very low pain threshold) and allodynia (amplified response to painful stimuli).

The treatment of fibromyalgia is symptomatic and the drugs only serve to reduce symptoms in some patients, in addition to the fact that these available treatments (antidepressants, pain signal modulators, rescue analgesics, etc.) have many side effects.

The food supplement which is the object of this study, FibrofixPlus®, is made up of a combination of natural substances.

This is the reason why this observational study aims to improve symptoms caused by fibromyalgia in patients treated with FibrofixPlus®.

DETAILED DESCRIPTION:
Patients who meet the fibromyalgia criteria according to the definition of the American College of Rheumatology (ACR) in 1990 and 2010, with a minimum score of 4 on the Visual Analogue Scale (VAS) of Fatigue and Pain and without any treatment (anxiolytics, neuroleptics, antidepressants and/or narcotic analgesics) in a minimum of 4 weeks prior to the beginning of the study, with some exceptions, and who do not meet any of the exclusion criteria will be invited to participate in the study.

There are three study visits which are distributed throughout 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years.
* Meet the fibromyalgia criteria according to the definition of the American College of Rheumatology of 1990 and 2010.
* Minimum score of 4 on the Visual Analogue Scale (VAS) for Fatigue and Pain.
* Period prior to the start of the study of a minimum of 4 weeks without treatment with anxiolytics, neuroleptics, antidepressants and/or narcotic analgesics. The use of paracetamol up to 2 g/day is allowed, and tramadol 100 mg/8h maximum.

Exclusion Criteria:

* Current diagnosis of a psychiatric disorder other than major depressive disorder.
* Pain caused by a traumatic or structural injury.
* Chronic inflammatory diseases.
* Autoimmune disease.
* Use of medications that may interfere with the assessment of pain improvement, including analgesics (with the exception stated in the inclusion criteria), antidepressants, anticonvulsants, or other medication taken to combat fibromyalgia, fatigue or pain.
* Rehabilitation with therapeutic intent.
* Intent to apply or current disability application process.
* Natural therapies (homeotherapy, acupuncture, food, etc.) to improve fibromyalgia.
* Hypersensitivity to the active principles or to any of the excipients of the products included in the study.
* Pregnancy.
* Breastfeeding.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women with fibromyalgia in primary care clinic.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
Symptomatic change of fibromyalgia through the Fibromyalgia Impact Questionnaire (s-FIQ), after taking the FibrofixPlus® food supplement, for 8 weeks. | From Visit 0, and at each visit (Visit 1 or 4 weeks after Visit 0; and Visit 2 or 8 weeks after Visit 0).
  To assess the magnitude of the symptomatic improvement by measuring the results to questions of the Fibromyalgia Impact Questionnaire (s-FIQ). This questionnaire scores from 0 to 100, being 0 the best quality of life and functional capacity, and 100 is the worst result.

SECONDARY OUTCOMES:
Rate of safety episodes. | Visit 1 to Visit 2, up to 4 weeks.
  All episodes will be recorded, whether considered minor or serious, food supplement-related or not.
Change of fatigue symptom through the Visual Analogue Scale (VAS). | From Visit 0, and at each visit (Visit 1 or 4 weeks after Visit 0; and Visit 2 or 8 weeks after Visit 0).
  To assess the fatigue symptom by the completion of the Visual Analogue Scale (VAS).
  The VAS scores from 0 to 10, being 0 the best outcome (without fatigue) and 10 the worst outcome (maximum fatigue).
Change of fatigue symptom through the Symptom Severity Score (SS Score). | From Visit 0, and at each visit (Visit 1 or 4 weeks after Visit 0; and Visit 2 or 8 weeks after Visit 0).
  To assess the fatigue symptom by the completion of the Symptom Severity Score (SS Score).
  The SS Score has a scoring from 0 to 12, being 0 the best outcome (without fatigue) and 12 the worst outcome (maximum fatigue).
Change of pain symptom through the Visual Analogue Scale (VAS). | From Visit 0, and at each visit (Visit 1 or 4 weeks after Visit 0; and Visit 2 or 8 weeks after Visit 0).
  To assess the pain symptom by the completion of the Visual Analogue Scale (VAS).
  The VAS scores from 0 to 10, being 0 the best outcome (without fatigue) and 10 the worst outcome (maximum fatigue).
Change of pain symptom through the Widespread Pain Index (WPI). | From Visit 0, and at each visit (Visit 1 or 4 weeks after Visit 0; and Visit 2 or 8 weeks after Visit 0).
  To assess the pain symptom by the completion of the Widespread Pain Index (WPI).
  The WPI scores from 0 to 19, being the highest result the worst outcome as defined by the number of body areas with pain.
Change of pain symptom through the Symptom Severity Score (SS Score). | From Visit 0, and at each visit (Visit 1 or 4 weeks after Visit 0; and Visit 2 or 8 weeks after Visit 0).
  To assess the pain symptom by the completion of the Symptom Severity Score (SS Score).
  The SS Score has a scoring from 0 to 12, being 0 the best outcome and 12 the worst outcome.
Change of the sleep quality through the Pittsburgh Sleep Quality Index (PSQI). | From Visit 0, and at each visit (Visit 1 or 4 weeks after Visit 0; and Visit 2 or 8 weeks after Visit 0).
  To assess the sleep quality by the completion of the Pittsburgh Sleep Quality Index (PSQI).
  The PSQI has a scoring from 0 to 21, being 0 the best outcome with no difficulties to sleep.
Change of the sleep quality through the Symptom Severity Score (SS Score). | From Visit 0, and at each visit (Visit 1 or 4 weeks after Visit 0; and Visit 2 or 8 weeks after Visit 0).
  To assess the sleep quality by the completion of the Symptom Severity Score (SS Score).
  The SS Score has a scoring from 0 to 12, being 0 the best outcome and 12 the worst outcome.
Change on the functional impairment through the questionnaire Clinical Global Impressions (CGI). | From Visit 0, and at each visit (Visit 1 or 4 weeks after Visit 0; and Visit 2 or 8 weeks after Visit 0).
  To assess the functional impairment by the completion of the Clinical Global Impressions (CGI).
  The CGI has a scoring from 0 to 7, being 0 "not assessed" and 1 "normal or not ill" and 7 "extremely ill".
Change on the functional impairment through the questionnaire Short Form-36 Questionnaire (SF-36). | At Visit 0 and at Visit 2, or 8 weeks after Visit 0.
  To assess the functional impairment by the completion of the Short Form-36 Questionnaire (SF-36).
  The SF-36 has several questions so when the scoring is higher, better is the health status. The global score is between 0 and 100, being 0 the worst and 100 the best health status.
Change on the quality of life through the questionnaire Clinical Global Impressions (CGI). | From Visit 0, and at each visit (Visit 1 or 4 weeks after Visit 0; and Visit 2 or 8 weeks after Visit 0).
  To assess the quality of life by the completion of the questionnaire CGI. The CGI has a scoring from 0 to 7, being 0 "not assessed" and 1 "normal or not ill" and 7 "extremely ill".
Change on the quality of life through the questionnaire Hospital Anxiety and Depression Scale (HADS). | At Visit 0 and at Visit 2, or 8 weeks after Visit 0.
  To assess the quality of life by the completion of the HADS. The HADS has a maximum score of 21, which indicates a severe or worse status.
Change on the quality of life through the questionnaire Short Form-36. | At Visit 0 and at Visit 2, or 8 weeks after Visit 0.
  To assess the quality of life by the completion of the Short Form-36 Questionnaire (SF-36).
  The SF-36 has several questions so when the scoring is higher, better is the health status. The global score is between 0 and 100, being 0 the worst and 100 the best health status.

CONTACTS AND LOCATIONS:
Overall Officials: Rodríguez Araya, Dr, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided